CLINICAL TRIAL: NCT05402371
Title: A Phase 2B, Randomized, Multi-Center, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Rencofilstat in Adult Subjects With Nonalcoholic Steatohepatitis and Advanced Liver Fibrosis
Brief Title: A Study to Evaluate the Efficacy and Safety of Rencofilstat in Subjects With NASH and Advanced Liver Fibrosis
Acronym: ASCEND
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hepion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEPA-CRV431-207
Record Dates: First submitted 2022-05-20; First posted 2022-06-02 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Nonalcoholic Steatohepatitis (NASH); Fibrosis, Liver; NAFLD
Keywords: Nonalcoholic Steatohepatitis; NAFLD; NASH; liver fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — CRV-431

STUDY DESIGN:
Intervention Model Description: blinded, placebo controlled, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A: Rencofilstat 75 mg (Experimental): Eighty-four (84) biopsy-proven NASH F2/F3 subjects to complete study on Rencofilstat 75 mg daily.
  Interventions: Drug: Rencofilstat
- Cohort B: Rencofilstat 150 mg (Experimental): Eighty-four (84) biopsy-proven NASH F2/F3 subjects to complete study on Rencofilstat 150 mg daily.
  Interventions: Drug: Rencofilstat
- Cohort C: Rencofilstat 225 mg (Experimental): Eighty-four (84) biopsy-proven NASH F2/F3 subjects to complete study on Rencofilstat 225 mg daily.
  Interventions: Drug: Rencofilstat
- Cohort D: Placebo (Placebo Comparator): Eighty-four (84) biopsy-proven NASH F2 / F3 subjects to complete study on matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rencofilstat — Rencofilstat soft gel capsule
  Other Names: CRV431
  Arms: Cohort A: Rencofilstat 75 mg; Cohort B: Rencofilstat 150 mg; Cohort C: Rencofilstat 225 mg
Drug: Placebo — placebo soft gel capsule
  Arms: Cohort D: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-dosing, multi-center study to evaluate the efficacy and safety of Rencofilstat as evidenced by histopathological improvements in fibrosis in adult NASH subjects with F2 or F3 fibrosis (NASH CRN system). Antifibrotic biomarker activity will be evaluated on an exploratory basis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-dosing, multi-center study to evaluate the efficacy and safety of Rencofilstat as evidenced by histopathological improvements in fibrosis in adult NASH subjects with F2 or F3 fibrosis (NASH CRN system). Antifibrotic biomarker activity will be evaluated on an exploratory basis.

This study consists of 3 phases: (i) Screening and Randomization; (ii) treatment; and (iii) follow up. During Screening, each subject will provide informed consent prior to starting any study specific procedures. The randomization of the F2/F3 NASH subjects will be performed in a 1:1:1:1 ratio between Rencofilstat 75mg, Rencofilstat 150mg, Rencofilstat 225mg, and matching placebo. Subjects will be stratified by presence or absence of Type 2 diabetes, fibrosis stage and a maximum of 34 F2 subjects in each cohort.

ELIGIBILITY:
Inclusion Criteria Subjects must fulfill all the following inclusion criteria to be eligible for participation in the study.

1. Male or female between 18 and 75 years of age (inclusive).
2. Capable of giving written informed consent and able to effectively communicate with the investigator and study personnel.
3. Histologic evidence of NASH based on central readings of the screening biopsy obtained no more than 6 months before Screening defined by presence of all 3 key histological features, Nonalcoholic Fatty Liver Disease Activity Score (NAS) ≥ 4 with at least 1 point each in lobular inflammation and hepatocyte ballooning.

   a. Historical biopsy may be substituted for Screening biopsy to determine eligibility if the following are met: i. Historical biopsy was obtained no more than 180 ± 5 days prior to the first day of Screening.

   ii. Hepatic tissue or slides are available for central histologic evaluation. iii. No new therapeutic intervention for NASH was made 90 days prior to screening (e.g., obeticholic acid, vitamin E ≥ 400 IU/day, pioglitazone, incretins [e.g., liraglutide, semaglutide], sodium-glucose cotransporter-2 [SGLT2] inhibitors).

   iv. Subjects must have been metabolically stable since the biopsy (no significant weight loss ≥ 7% of body weight, no major deterioration of glycemic control, and no introduction of new or investigational drugs for the treatment of Type 2 Diabetes).
4. Histologic liver fibrosis stage 2 or 3 as defined by the Nonalcoholic Steatohepatitis Clinical Research Network (NASH CRN) scoring of liver fibrosis based on central reading of the Screening biopsy (refer to criteria 4a regarding use of a historical biopsy as a substitute for the Screening biopsy).
5. Blood pressure up to 160/100 mmHg; potential subjects who meet other eligibility requirements, but who have out of range blood pressure measurements deemed to be not clinically significant by the investigator, may still be considered for study inclusion.

Exclusion Criteria Subjects who meet any of the following criteria prior to the first dose of study drug are not eligible for randomization.

1. Pregnant or breastfeeding or planning to become pregnant during the study period.
2. Known allergy to Rencofilstat, cyclosporine, or any of their inactive ingredients.
3. Positive test for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCVAb) or human immunodeficiency virus antibodies (HIVAb). If HCVAb test is positive, then an HCV-RNA test will be performed. If this test is negative, the subject is allowed to participate in the study, as long as the subject meets all other inclusion criteria and has never been treated for HCV or was treated >2 years ago and achieved a sustained virologic response at that time.
4. Subjects with suspected and symptomatic severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection identified prior to first dose.
5. Subjects with a history of clinically significant acute cardiac events within 30 days prior to Screening such as stroke, transient ischemic attack, or coronary heart disease (angina pectoris requiring therapy, myocardial infarction, revascularization procedures with left ventricular ejection fraction [LVEF] <50% as determined by previous echocardiography or multiple gated acquisition [MUGA] scan).
6. Subjects with uncontrolled or unstable cardiac arrhythmias:

   1. Severe conduction disturbance (e.g., second-degree or third-degree AV block).
   2. History of congenital long QT syndrome, congenital short QT syndrome, Torsades de Pointes, or Wolff Parkinson White syndrome.
7. Subjects with transaminases >5 x upper limit of normal (ULN).
8. Subjects with ALP >2 x ULN.
9. Subjects with total serum bilirubin >1.5 x ULN.
10. Subjects with a platelet count <100,000/mm3.
11. Subjects with an INR ≥ 1.3 in the absence of anticoagulants.
12. Subjects with albumin <3.5 g/dL.
13. Model for End-Stage Liver Disease (MELD) score >12, unless due to an alternate etiology such as therapeutic anticoagulation.
14. Current or previous (within the past 6 months) Child-Pugh (CP) score ≥ 7 for F2 or F3 subjects, unless due to an alternative etiology such as Gilbert's syndrome or therapeutic anticoagulation.
15. An estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 (calculated by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] method).
16. Subjects with hemoglobin A1c (HbA1c) >9.5%.
17. Subjects with any history or presence of decompensated cirrhosis including ascites, hepatic encephalopathy or variceal bleeding.
18. Other well documented causes of chronic liver disease according to standard diagnostic procedures including, but not restricted to:

    1. Suspicion of drug-induced liver disease.
    2. Alcoholic liver disease.
    3. Autoimmune hepatitis.
    4. Wilson's disease.
    5. Primary biliary cholangitis, primary sclerosing cholangitis.
    6. Genetic hemochromatosis (Homozygosity for C282Y or C282Y/H63D compound heterozygote).
    7. Known or suspected hepatocellular carcinoma (HCC).
    8. History or planned liver transplant.
    9. Clinical evidence of portal hypertension such as esophageal varices, ascites, history of hepatic encephalopathy, or splenomegaly.
19. History of hepatic decompensating events or subjects who develop manifestations of hepatic decompensation between screening and enrollment should not be randomized, inclusive of new or worsening jaundice and ascites, new esophageal varices, etc.
20. Subjects with Type 2 diabetes who have recent (< 3 months) changes in medication class or dose of the following antidiabetic medications: Glucagon-like-peptide-1 (GLP-1) receptor agonist, dipeptidyl peptidase-4 (DPP-4) inhibitor, sodium/glucose cotransporter 2 (SGLT2) inhibitor, thiazolidinediones (TZD).
21. Received an investigational drug or investigational vaccine or used an investigational medical device within 60 days prior to first dose of study drug.
22. Received any investigation products being evaluated for the treatment of liver fibrosis or NASH in the 6 months prior to the Screening liver biopsy.
23. Inability to undergo MRE procedure due to unremovable metal or foreign object(s) or contraindication for any other reason including but not limited to pacemaker, shrapnel injury, extensive tattoos, severe claustrophobia, ear (cochlea) implant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with improvement in fibrosis by at least 1 stage (NASH CRN system) OR NASH resolution without worsening of fibrosis. | dosing period of 1 year with 1 month observation and follow up period
  Efficacy

SECONDARY OUTCOMES:
Proportion of subjects with improvement in fibrosis by at least 1 stage (NASH CRN system), regardless of effect on NASH. | dosing period of 1 year with 1 month observation and follow up period
  Efficacy
Proportion of subjects with improvement in fibrosis by at least 2 stages (NASH CRN system), regardless of effect on NASH. | dosing period of 1 year with 1 month observation and follow up period
  Efficacy
Proportion of subjects with improvement in fibrosis by at least 2 stages (NASH CRN system) AND no worsening of NASH. | dosing period of 1 year with 1 month observation and follow up period
  Efficacy
Change from baseline in ALT. | dosing period of 1 year with 1 month observation and follow up period
  Efficacy
Change from baseline in AST. | dosing period of 1 year with 1 month observation and follow up period
  Efficacy
Change from baseline in Pro-C3, type III collagen neo-epitopes. | dosing period of 1 year with 1 month observation and follow up period
  Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Harrison, MD, Principal Investigator — Pinnacle Clinical Research
Locations (41):
- United States (39):
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Arizona Liver Health-Chandler, Chandler, Arizona
  - Arizona Liver Health, Peoria, Arizona
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - Arizona Liver Health-Tuscon, Tucson, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - National Research Institute, Huntington Park, California
  - National Research Institute, Los Angeles, California
  - National Research Institute, Panorama City, California
  - National Research Institute, Santa Ana, California
  - Synergy Healthcare, LLC, Bradenton, Florida
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - Top Medical Research, Inc., Cutler Bay, Florida
  - Integrity Clinical Research, LLC, Doral, Florida
  - Evolution Clinical Trials, Inc., Hialeah Gardens, Florida
  - Borland Groover Clinical Research, Jacksonville, Florida
  - Ocala GI Research, Lady Lake, Florida
  - Accel Research Sites-Lakeland CRU, Lakeland, Florida
  - Future Care Solutions, LLC, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - United Reseach Group, Miami, Florida
  - Omega Research Consultants, LLC, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Covenant Research and Clinics, Sarasota, Florida
  - Southeast Clinical Research Center, Dalton, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Digestive Research Alliance of Michiana, LLC, South Bend, Indiana
  - Delta Research Partners, Bastrop, Louisiana
  - Mid-Atlantic GI Research, LLC, Greenbelt, Maryland
  - AIG Digestive Disease Research, LLC, Florham Park, New Jersey
  - Pinnacle Clinical Research-Austin, Austin, Texas
  - South Texas Research Institute, Brownsville, Texas
  - South Texas Research Institute, Edinburg, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Pinnacle Clinical Research-San Antonio, San Antonio, Texas
  - Bon Secours Liver Institute of Hampton Roads, Newport News, Virginia
  - GI Select Health Research, LLC, Richmond, Virginia
  - Velocity Clinical Spokane, Spokane, Washington
- Hopital du Haut Leveque, Pessac, France
- Centro de Investigacion y Gastroenterologia SC, Mexico City, Mexico